CLINICAL TRIAL: NCT00558805
Title: Family Intervention for Suicidal Youth: Emergency Care
Acronym: FISP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 921708
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-10

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted | interventions — interleukin-24

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Usual Care + Family Intervention for Suicide Prevention (FISP)
  Interventions: Behavioral: FISP + Usual Care
- 2 (Other): Usual Care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: FISP + Usual Care
  Arms: 1
Behavioral: Usual Care
  Arms: 2

SUMMARY:
This project evaluates a brief intervention in the emergency department (ED) for adolescents presenting with suicide attempts. The intervention aims to capitalize on the opportunity offered by the ED visit to deliver an effective intervention, improve adherence to follow-up care, decrease the risk of repeat suicide attempts, and improve clinical and functioning outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 years
* Suicidal patient presenting to Emergency Department

Exclusion Criteria:

* Acute psychosis/symptoms that impede consent/assessment
* No parent/guardian to consent (youth <18)
* Youth not English-speaking
* Parents/guardians not English or Spanish-speaking.

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Joan R Asarnow, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Emergency Medical Center, Los Angeles, California
  - Los Angeles County Harbor-UCLA Medical Center, Los Angeles, California

REFERENCES:
- [Derived] Asarnow JR, Baraff LJ, Berk M, Grob CS, Devich-Navarro M, Suddath R, Piacentini JC, Rotheram-Borus MJ, Cohen D, Tang L. An emergency department intervention for linking pediatric suicidal patients to follow-up mental health treatment. Psychiatr Serv. 2011 Nov;62(11):1303-9. doi: 10.1176/ps.62.11.pss6211_1303. PMID 22211209